CLINICAL TRIAL: NCT03373474
Title: Comparison of Effectiveness Between Warm Acupuncture With Local-Distal Points Association and Local Distribution Points Association in Breast Cancer Related Lymphedema Patients: A Multicenter, Randomized, Controlled Clinical Trial
Brief Title: Warm Acupuncture for Breast Cancer Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin University of Traditional Chinese Medicine (Other)
Collaborators: National Basic Research Program, China (Other); Tianjin Medical University Cancer Institute and Hospital (Other); The Second Affiliated Hospital of Baotou Medical College (Other); Henan Provincial People's Hospital (Other); Qilu Hospital of Shandong University (Other); Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Yi Guo, The Dean of Acupuncture and Moxibustion College, Tianjin University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014CB543202-02
Record Dates: First submitted 2017-12-07; First posted 2017-12-14 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- local distribution points association (Experimental): Participants will receive warm acupuncture with the local distribution acupoints association on the affected arm only.
  Interventions: Other: local distribution points association
- local-distal points association (Experimental): Participants will receive warm acupuncture with the local-distal acupoints association on the affected arm, unaffected arm, abdomen, and legs.
  Interventions: Other: local-distal points association
- waiting-list (No Intervention): Patients in the waiting-list group will not receive any acupuncture treatment during the study. However, for ethical consideration, 20 free acupuncture treatments will be offered after the study is completed.

INTERVENTIONS:
Other: local distribution points association — Participants will receive acupuncture treatments using the local points set plus the local-addition points set (local distribution association) described below. Warming acupuncture will be applied at HT2, LI11, and TE9 if permitted.
  Local points set: TE5, LI11, TE9, HT3, TE13, and Xiajiquan on the affected arm. Local-addition points set: LU5, PC3, SI7, TE4, TE3, HT2, TE10, LI15, and 2 other points according to the symptom on the affected arm.
  Arms: local distribution points association
Other: local-distal points association — Participants will receive acupuncture treatments using the local points set plus the distal points set (local-distal association) described below. Warming acupuncture will be applied similarly to the local distribution group, with the addition of Ren6, Ren9, bilateral SP9, and LI11 on the unaffected arm.
  Local points set: TE5, LI11, TE9, HT3, TE13, and Xiajiquan on the affected arm. Distal points set: TE5, LI11, HT3, TE13 on the unaffected arm; CV4, CV6, CV9, CV12, bilateral SP6 and SP9.
  Arms: local-distal points association

SUMMARY:
The purpose of this study is to clarify whether local-distal point association is more effective than local point association by warm acupuncture in the management of breast cancer related lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months after breast cancer surgery and presents with persistent breast cancer related upper extremity lymphedema for at least 3 months. Upper extremity lymphedema is defined as more than 2cm circumference difference or 5% volume difference between the affected and unaffected arms.
* Stage II or III lymphedema according to the 2016 consensus by the international society of lymphology.
* Karnofsky Performance Score (KPS) ≥ 70
* Men or women aged 18 to 80 years
* Out-patients
* Estimated life expectancy > 6 months

Exclusion Criteria:

* Bilateral breast cancer related lymphedema
* Taking diuretic
* History of primary lymphedema
* A diagnosis of severe heart, liver, kidney or hematologic disease
* Edema caused by upper extremity disability or other conditions such as heart failure, kidney disease or malnutrition
* Have hypoproteinemia
* Inflammation, scar, or trauma at the site of operation, or other active skin infections
* Unable to self-care, had a history of psychological disorders, or unable to communicate
* Received lymphedema treatment within the past 1 month
* Pregnancy or breastfeeding
* The presence of electronic medical device implants
* Deny to sign the informed written consent, or unwilling to conform to randomization
* Participation in other clinical trials during the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-12-26 (Actual)

PRIMARY OUTCOMES:
Upper extremity circumference | 80 weeks
  Various assessment methods are available but circumference measure is simple, convenient with low cost, and reliable. Therefore, the primary outcome measures will be the mean change in inter-limb circumference difference from baseline to the end of the 8-week intervention. The circumference will be measured by the measurement tape (Gulick Attachment, Baseline, America) at the wrist crease, 10 cm above the wrist crease, elbow crease, 10 cm above the elbow crease, where the lymphedema is most severe and its corresponding location on the unaffected limb.

SECONDARY OUTCOMES:
Upper extremity volume | 80 weeks
  Volume measurement is also commonly used for the evaluation of lymphedema and the mean change in inter-limb volume difference from baseline to the end of the 8-week intervention will be included as the second primary outcome measure. The volume of the affected and unaffected limb will be measured by the volumetric measuring device (Baseline, America) using the water displacement method, which is considered as the most reliable method for volume measurements.
Common terminology criteria for adverse events (CTCAE 4.03) - edema limbs criteria | 80 weeks
  Common terminology criteria for adverse events (CTCAE 4.03) will be used to grade the severity of swelling using the edema limbs criteria. A grading of mild, moderate or severe swelling will be assessed based on the inter-limb circumference or volume discrepancy, anatomic architecture, appearance, or activities of daily living. The CTCAE 4.03 will allow us to evaluate the clinical significance of circumference change.
Stages of lymphedema from the international society of lymphology | 80 weeks
  Stages of lymphedema from the international society of lymphology will be used to grade the severity of lymphedema. Staging of 0, I, II, or III will be assessed based on severity of swelling, ability to reduce swelling by elevation, and skin changes.
The Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure | 80 weeks
  Disabilities of the arm, shoulder, and hand (DASH) is a scale consists of two concepts: functional status (part A) and symptoms (part B) respectively. The functional status part is further divided into three dimensions: physical, social, and psychological. The total score of the DASH ranges from 0 to 100 with higher scores representing worse symptoms and function. The DASH has good validity and responsiveness and it is recommended to assess upper extremity function in breast cancer survivors. The validated Chinese version of the DASH will be used in this study.
The MOS 36-Item Short-Form Health Survey (SF-36) | 80 weeks
  The medical outcome study 36-item short-form health survey (SF-36) is a commonly used instrument to assess quality of life that has good validity. The SF-36 includes the following eight concepts: physical functioning, role limitations due to physical problems, social functioning, bodily pain, general mental health, role limitations due to emotional problems, vitality, and general health perception. The validated Chinese version of the SF-36 will be used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: XingFang Pan, Principal Investigator — Baokang Hospital Affiliated to Tianjin University of Traditional Chinese Medicine
Locations (1):
- Baokang Hospital Affiliated to Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Yeh CH, Zhao TY, Zhao MD, Wu Y, Guo YM, Pan ZY, Dong RW, Chen B, Wang B, Wen JR, Li D, Guo Y, Pan XF. Comparison of effectiveness between warm acupuncture with local-distal points combination and local distribution points combination in breast cancer-related lymphedema patients: a study protocol for a multicenter, randomized, controlled clinical trial. Trials. 2019 Jul 5;20(1):403. doi: 10.1186/s13063-019-3491-4. PMID 31277678